CLINICAL TRIAL: NCT06853756
Title: Gastric Insufflation Volume Using I-gel Versus Ambu AuraGain in Pediatric Patients Undergoing Elective Orthopedic Operations Under General Anesthesia: a Prospective Randomized Trial
Brief Title: Gastric Insufflation Volume Using I-gel Versus Ambu AuraGain in Pediatric Patients Undergoing Elective Orthopedic Operations Under General Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Nabil Farahat, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36264MS287/8/23
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Gastric Insufflation; I-gel; Ambu AuraGain; Pediatric; Orthopedic Operations; General Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambu Auragain group (Experimental): Ambu Auragain was inserted after induction.
  Interventions: Device: Ambu Auragain
- I-gel group (Experimental): The I-gel device was inserted after induction.
  Interventions: Device: I-gel

INTERVENTIONS:
Device: Ambu Auragain — Ambu Auragain was inserted after induction.
  Arms: Ambu Auragain group
Device: I-gel — The I-gel device was inserted after induction.
  Arms: I-gel group

SUMMARY:
Our study aimed to compare the gastric insufflation volume between Ambu AuraGain and i-gel and its relationship with the oropharyngeal sealing pressure and the incidence of postoperative complications in generally anesthetized controlled-ventilated pediatric patients undergoing elective orthopedic operations.

DETAILED DESCRIPTION:
Supraglottic Airway Devices (SADs) refer to a wide range of medical devices that can act as a passageway for oxygenation, ventilation, and administration of anesthetic gases and may be deemed an alternative to Endotracheal Tubes (ETTs).

Oropharyngeal sealing pressure (OLP) provides insight into the risk of gastric insufflation and aspiration risk. It is considered a measure of adequate performance and successful placement based on the premise that the SAD is sited properly in the hypopharynx after blind placements, and it is a useful comparator between SADs.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 2 to 12 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I and II.
* Scheduled for elective orthopedic operations in a supine position under general anesthesia.

Exclusion Criteria:

* Patients with a known history of gastro-oesophageal reflux disorders.
* Full Stomach.
* Anticipated difficult mask ventilation or intubation.
* Body mass index "BMI" exceeding 20% of the ideal.
* A history of chest problems.
* History of the gastrointestinal tract or thoracic surgeries.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-03-27 (Estimated); Study Completion 2025-03-27 (Estimated)

PRIMARY OUTCOMES:
Gastric antrum cross-sectional area (CSA) | At the end of surgery before supraglottic airway devices removal (5 min)
  Gastric antrum cross-sectional area (CSA) was measured before induction of general anesthesia, before supraglottic airway devices (SAD) insertion, after Ryle's tube insertion, and at the end of surgery before SAD removal.

SECONDARY OUTCOMES:
Oropharyngeal leak pressure | Intraoperatively
  Oropharyngeal leak pressure was determined after confirmation of adequate device insertion and secure taping by closing the adjustable pressure-limiting (APL) valve with a fresh gas flow of 3 l/min and observing the airway pressure at which equilibrium was attained in the aneroid manometer (airway pressure was not allowed to exceed 40cmH2O) or when there was audible air leak from the throat which was auscultated in the neck with a stethoscope placed just beside the thyroid cartilage.
Time of insertion of supraglottic airway devices | Intraoperatively
  Insertion time was measured in seconds and counted from the time of opening the jaw to the appearance of the capnography waveform.
Number of attempts for insertion | Intraoperatively
  Three insertion attempts were allowed. Each 'attempt' was defined as reinsertion of the airway device into the mouth. Insertion failure of the device was defined as greater than three unsuccessful attempts or if the entire process of insertion exceeded 120 seconds.
Incidence of postoperative complications | 24 hours postoperatively
  Incidence of postoperative complications such as mucosal injury, laryngeal spasm, hoarseness, nausea and vomiting were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.